CLINICAL TRIAL: NCT05925751
Title: An Integration of a Computed Tomography/Positron Emission Tomography/Whole Slide Image (CT/PET/WSI) Based Deep Learning Signature for Predicting Complete Pathological Response to Neoadjuvant Chemoimmunotherapy in Non-small Cell Lung Cancer: A Multicenter Study
Brief Title: Deep Learning Signature for Predicting Complete Pathological Response to Neoadjuvant Chemoimmunotherapy in Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Ningbo No.2 Hospital (Other); Zunyi Medical College (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: DLCPR
Record Dates: First submitted 2023-05-12; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer; Neoadjuvant Chemoimmunotherapy; Complete Pathological Response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT/PET/WSI-based Deep Learning Signature — CT/PET/WSI-based Deep Learning Signature for Predicting Complete Pathological Response to Neoadjuvant Chemoimmunotherapy in Non-small Cell Lung Cancer

SUMMARY:
The purpose of this study is to evaluate the performance of a CT/PET/ WSI-based deep learning signature for predicting complete pathological response to neoadjuvant chemoimmunotherapy in non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 20-75 years;
2. Patients who underwent curative surgery after neoadjuvant chemoimmunotherapy for NSCLC;
3. Obtained written informed consent.

Exclusion Criteria:

1. Missing image data;
2. Pathological N3 disease.

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Resected Stage I-III NSCLC following neoadjuvant chemoimmunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve | 2023.5.1-2023.10.31
  The area under the receiver operating characteristic curve (ROC) of the deep learning model in predicting complete pathological response (CPR). CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.

SECONDARY OUTCOMES:
Sensitivity | 2023.5.1-2023.10.31
  The sensitivity of the deep learning model in predicting complete pathological response. CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.

OTHER OUTCOMES:
Specificity | 2023.5.1-2023.10.31
  The specificity of the deep learning model in predicting complete pathological response. CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.
Positive predictive value | 2023.5.1-2023.10.31
  The positive predictive value of the deep learning model in predicting complete pathological response. CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.
Negative predictive value | 2023.5.1-2023.10.31
  The negative predictive value of the deep learning model in predicting complete pathological response. CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.
Accuracy | 2023.5.1-2023.10.31
  The accuracy of the deep learning model in predicting complete pathological response. CPR was defined as no residual tumor in both resected primary tumor and lymph nodes. Patients with non-small cell lung cancer receiving neoadjuvant chemoimmunotherapy will achieve either CPR or non-CPR, which can be confirmed by pathological examination after surgical resection. And the model will output the predictive value (CPR/non-CPR) for each patient receiving neoadjuvant chemoimmunotherapy.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ningbo HwaMei Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No